CLINICAL TRIAL: NCT03631342
Title: Comparison Between Different Ventilator Hyperinflation Maneuvers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brazilian Institute of Higher Education of Censa (Other)
Responsible Party: Principal Investigator, Luciano Matos Chicayban, Principal Investigator, Brazilian Institute of Higher Education of Censa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: VHI Modality
Record Dates: First submitted 2018-08-06; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Infections, Respiratory; Ventilator Associated Pneumonia
Keywords: Ventilator Hyperinflation; Physical Therapy; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: In order to perform both interventions, the patients were placed in dorsal decubitus with a head elevated at 45 ° and submitted to closed tracheal aspiration, according to the recommendations of the American Association for Respiratory Care. In addition, the bacteriological filter was changed, the cuff pressure was increased and the presence of leaks in the mechanical fan circuits was verified.
  All patients underwent five hyperinflation maneuvers, the order being determined by randomization. Controlled volume ventilation (VCV) at a constant flow rate of 20 Lpm (VCV-20) and 40 Lpm (VCV-40), controlled pressure ventilation (VCV-40) was performed for 2 minutes at 10 minute intervals. PCV), pressure-controlled ventilation associated with inspiratory time adjustment (PCV + Tins) and pressure-supported ventilation (PSV). PEEP and FiO2 were maintained throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VCV20 (Experimental): Volume-controlled ventilation mode under constant flow of 20 Lpm. The inspired volume was progressively increased until the maximum pressure reached 40cmH2O.
  Interventions: Other: VCV20
- VCV40 (Experimental): Volume controlled ventilation mode under constant flow of 40 Lpm. The inspired volume was progressively increased until the maximum pressure reached 40cmH2O.
  Interventions: Other: VCV40
- PCV (Experimental): Pressure controlled ventilation mode, inspiratory time of 1 second. The inspiratory pressure was increased every 5 cmH2O, until reaching the maximum pressure of 40 cmH2O.
  Interventions: Other: PCV
- PCV+Tins (Experimental): Pressure controlled ventilation mode and inspiratory pressure was increased every 5cmH2O, until the maximum pressure of 40 cmH2O was reached. The inspiratory time was gradually increased until the inspiratory flow reached the baseline. Concomitantly, the respiratory rate was decreased to allow the expiratory flow also to reach the baseline, to avoid self-PEEP.
  Interventions: Other: PCV+Tins
- PSV (Experimental): Pressure support ventilation mode, with progressive increases of 5 cmH2O at inspiratory pressure, until reaching Pmax of 40 cmH2O. The expiratory sensitivity was adjusted by 25% for all patients.
  Interventions: Other: PSV

INTERVENTIONS:
Other: VCV20 — controlled volume ventilation mode under constant flow of 20 Lpm. The inspired volume was progressively increased until the Pmax reached 40cmH2O.
  Arms: VCV20
Other: VCV40 — volume controlled ventilation mode under constant flow of 40 Lpm. The inspired volume was progressively increased until the Pmax reached 40cmH2O.
  Arms: VCV40
Other: PCV — controlled ventilation mode, 1 second inspiratory time. The inspiratory pressure was increased every 5 cmH2O, until reaching the maximum pressure of 40 cmH2O.
  Arms: PCV
Other: PCV+Tins — controlled ventilation and inspiratory pressure was increased every 5 cmH2O until the maximum pressure was 40 cmH2O. The inspiratory time was gradually increased until the inspiratory flow reached the baseline. Concomitantly, the respiratory rate was decreased to allow the expiratory flow also to reach the baseline, to avoid self-PEEP.
  Arms: PCV+Tins
Other: PSV — ventilatory mode with pressure support, with progressive increases of 5 cmH2O at inspiratory pressure, until reaching Pmax of 40 cmH2O. The expiratory sensitivity was adjusted by 25% for all patients.
  Arms: PSV

SUMMARY:
The hyperinflation ventilator was performed in different modalities and ventilatory adjustments, with total pressure of 40cmH2O. The inspiratory volume, inspiratory time, mean airway pressure, inspiratory and expiratory flow, and bias flow were evaluated.

DETAILED DESCRIPTION:
PURPOSE: To compare different ways of applying ventilator hyperinflation. METHODS: A randomized crossover clinical trial was performed with 30 patients (66.5 ± 17.3 years) with hypersecretion. The ventilator hyperinflation was performed in five ventilatory modalities for five minutes, with an interval of 2 hours, the order being determined by randomization: controlled ventilation at volume (VCV) with constant flow of 20 (VCV20) Lpm and 40 Lpm (VCV40), controlled ventilation pressure ventilation (PCV), controlled pressure ventilation associated with inspiratory time adjustment (PCV + Tins) and support pressure ventilation (PSV). In VCV mode, the volume was increased every 50mL, until reaching a maximum pressure of 40cmH2O. In the pressure controlled modes, the inspiratory pressure was increased every 5 cmH2O until the total pressure reached 40 cmH2O. The inspiratory time was adjusted so that the inspiratory flow reached the baseline. The following variables were evaluated: tidal volume, inspiratory time (Tins), mean airway pressure (Pmean), peak inspiratory flow (PIFR) and expiratory flow (PEFR), PIFR / PEFR and Bias Flow (PEFR-PIFR).

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary infection
* Mechanically ventilated for more than 96 hours through pressure-assisted ventilation (PSV) or pressure-controlled ventilation (PCV)
* Static compliance between 30 and 70 mL/cmH2O
* PEEP between 5 and 8 cmH2O.

Exclusion Criteria:

* Hemodynamic instability
* Non-drained pleural effusion or pneumothorax
* Intracranial hypertension
* Bronchospasm
* Adult respiratory distress syndrome (ARDS)
* Decompensated congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Inspiratory Volume | Five minutes after the onset of intervention
  Inspiratory volume reached in each mode of ventilator hyperinflation, under a maximum pressure of 40cmH2O
Inspiratory time | Five minutes after the onset of intervention
  inspiratory time necessary for the inspiratory flow to reach the baseline or according to the settings of each modality
Mean Pressure | Five minutes after the onset of intervention
  airway mean pressure measured on the mechanical ventilator in 2 cycles
Peak Expiratory Flow | Five minutes after the onset of intervention
  maximal expiratory flow in 2 cycles
Peak Inspiratory Flow | Five minutes after the onset of intervention
  Maximal inspiratory flow in 2 cycles
PIFR/PEFR | Five minutes after the onset of intervention
  Peak inspiratory to expiratory flow ratio
Bias Flow | Five minutes after the onset of intervention
  Difference between peak inspiratory and expiratory flows

CONTACTS AND LOCATIONS:
Overall Officials: LUCIANO M CHICAYBAN, MSc, Principal Investigator — Brazilian Institute of Higher Education of Censa
Locations (1):
- Luciano M Chicayban, Campos dos Goytacazes, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No